CLINICAL TRIAL: NCT06086990
Title: Effects in Quality of Life of a Telemonitoring Platform Amongst Patients With Cancer: A Randomized Trial
Brief Title: Effects of Telemonitoring in Quality of Life Amongst Cancer Patients
Acronym: EQUALITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Collaborators: Centro para la Prevención y Control del Cáncer (CECAN), Santiago, Chile (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez Lomakin, Associate Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNAB-005
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Telemonitoring; Telemedicine; Symptoms and Signs; Quality of Life
Keywords: Telemonitoring; Internet; Web-based applications; Quality of Life; Smartphones; Cancer
MeSH Terms: conditions — Neoplasms; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a 1:1 fashion to receive the smartphone application or usual follow-up care.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome assessors, investigators and analysts will be kept unaware of treatment allocation. However, due to the characteristics of the intervention, it is not possible to mask participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring Platform (Experimental): Patients assigned to the active intervention group will have access to a smartphone application named "Contigo." This application is designed to identify signs and symptoms of oncology drug toxicity while providing educational content. It equips patients with the necessary tools to manage typical clinical situations associated with the diagnosis and treatment of their disease.
  Interventions: Device: Contigo Application
- Traditional Follow-Up (No Intervention): Individuals designated to the traditional follow-up group will undergo standard care, including in-person check-ups as determined by their attending physician.

INTERVENTIONS:
Device: Contigo Application — Contigo, a smartphone app, focuses on two main goals: monitoring cancer patients for early signs of drug toxicity and offering educational content to empower them in managing clinical challenges linked to their diagnosis and treatment. Monitoring involves patients inputting experiences via oncology-related questionnaires, with weekly checks for chemotherapy toxicity using a validated questionnaire (PRO-CTCAE). Severe cases trigger alerts, while milder ones receive educational guidance. Data collected is shared with healthcare providers. Educational content, backed by scientific evidence and expert collaboration, covers cancer-specific topics and healthcare processes to enhance patients' self-awareness and self-care practices.
  Arms: Telemonitoring Platform

SUMMARY:
This interventional study aims to explore the potential of a smartphone app, Contigo, in enhancing the quality of life for patients with various cancers compared to standard care. The investigators will asses effects on quality of life, depressive symptoms, and appointment adherence.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if utilizing a smartphone app for disease monitoring improves the self-reported quality of life using validated questionnaires in patients with diverse solid cancers compared to standard care. Secondary objectives focused on evaluating its impact on depressive symptoms and assessing adherence to in-person appointments. This study involves a randomized trial among patients recently diagnosed with specific forms of cancer and undergoing curative treatment at the UC Christus Cancer Center. The eligible participants, 80 adults with recent histologically confirmed cancer diagnoses, will be randomized to receive either the smartphone application (Contigo) or standard educational care. Randomization will be performed independently using an allocation sequence that will be kept concealed from clinical investigators. Contigo offers two primary functions: monitoring cancer patients and delivering educational content to aid patients in dealing with common clinical situations related to their disease. The study will assess outcomes such as quality of life changes, depressive symptom development, and adherence to in-person appointments. All analyses will be undertaken under the intention to treat principle by a statistician unaware of treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old).
* Recent histologically confirmed diagnosis (within the last 3 months) of bronchogenic, breast, gallbladder, gastric, colorectal, or prostate cancer in any of its forms.
* Awaiting initiation of curative intent treatment for the disease using any modality (radiation therapy, chemotherapy, immunotherapy, etc.) at the UC-Christus Cancer Center.
* Possession of a smartphone, regardless of its native operating system (iOS® or Android®).
* Willingness to sign an informed consent form to participate in the study.

Exclusion Criteria:

* Any form of sensory impairment preventing app usage.
* Cognitive impairment.
* Psychiatric pathology hindering app usage.
* Unwillingness to participate in the study.
* Concurrent participation in another clinical trial addressing healthcare technologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scores | 30, 60 and 90 days after randomization.
  Quality of Life as assessed by the EuroQol 5 Dimension (EQ-5D) questionnaire. The index score ranges from 0 to 1, with higher values indicating an overall better quality of life.

SECONDARY OUTCOMES:
Development of Symptoms of Depression | 30, 60 and 90 days after randomization.
  Development of symptoms of depression as evaluated by the Patient Health Questionnaire 9 (PHQ-9) scale. Scores can range from 0 to 27, with higher scores increasing the probability of depression.
Adherence to medical appointments | 90 days after randomization.
  Adherence to in-person medical appointments, as established by the attending physician of each participant. This outcome will be expressed as the proportion of visits attended by each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Nervi, MD, Study Chair — Pontificia Universidad Catolica de Chile; Manuel Gonzalez, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- UC Christus Cancer Centre, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized individual participant data, encompassing clinical characteristics and outcomes, will be accessible to fellow researchers upon reasonable request. This access can aid in conducting a systematic review on telemonitoring platforms for providing care to cancer patients.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Zarate V, Kind P, Valenzuela P, Vignau A, Olivares-Tirado P, Munoz A. Social valuation of EQ-5D health states: the Chilean case. Value Health. 2011 Dec;14(8):1135-41. doi: 10.1016/j.jval.2011.09.002. Epub 2011 Nov 6. PMID 22152184
- [Background] Sprave T, Gkika E, Verma V, Grosu AL, Stoian R. Patient reported outcomes based on EQ-5D-5L questionnaires in head and neck cancer patients: a real-world study. BMC Cancer. 2022 Nov 29;22(1):1236. doi: 10.1186/s12885-022-10346-4. PMID 36447175
- [Derived] Martinez F, Taramasco C, Espinoza M, Acevedo J, Goic C, Nervi B. Effects on Quality of Life of a Telemonitoring Platform amongst Patients with Cancer (EQUALITE): A Randomized Trial Protocol. Methods Protoc. 2024 Mar 15;7(2):24. doi: 10.3390/mps7020024. PMID 38525782
- See also: Center for Cancer Control and Prevention Website — https://cecan.cl/
- See also: UC Christus Cancer Center — https://www.ucchristus.cl/especialidades-y-servicios/especialidades/cancer-uc